CLINICAL TRIAL: NCT02274077
Title: Abdominal Wall Reconstruction: Postoperative Outcomes Using Transverse Abdominal Plane Anesthesia
Brief Title: Transverse Abdominal Plane Anesthesia for Abdominal Wall Reconstruction
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: funding for the study was terminated
Sponsor: Chester Mays (Other)
Responsible Party: Sponsor-Investigator, Chester Mays, Chief Resident, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSRB00042032
Record Dates: First submitted 2014-10-08; First posted 2014-10-24 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Hernia, Ventral
Keywords: length of stay; nausea; emesis; bowel function; pain scores; narcotic pain medication; post operative period
MeSH Terms: conditions — Hernia, Ventral; Nausea; Vomiting | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EXPAREL (Active Comparator): Bilateral, one time injections using 30ml of EXPAREL ((bupivacaine liposome injectable suspension) 1.3% ( 13.3mg/ml)) into the transverse abdominal plane at the time of abdominal component separation. A total of 60cc used with a Bupivacaine concentration of 0.44%.
  Interventions: Drug: EXPAREL
- Normal Saline (Placebo Comparator): Bilateral, one time injections of 30ml normal saline into the transverse abdominal plane at the time of abdominal component separation.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: EXPAREL
  Other Names: bupivacaine liposome injectable suspension
  Arms: EXPAREL
Drug: Normal Saline
  Arms: Normal Saline

SUMMARY:
The aim of this study is to evaluate the short-term postoperative outcomes in the abdominal wall reconstruction population using an intraoperative local anesthetic infusion. A prospective randomized double blind study of patients undergoing component separation will be performed in order to assess the following outcomes:

1. Length of Stay (LOS)
2. Return of bowel function
3. Narcotic pain medication requirements
4. Nausea and emesis
5. Pain scores

DETAILED DESCRIPTION:
One group will be the control group (group A) and the other will be the study group (group B). Neither patient nor physician will know which group they have been assigned. Informed consent will be obtained during pre-operative evaluation in the clinic prior to the day of surgery as stated above. Relevant medical history will be entered into a secure database. Information collected will include patient demographics, medical co-morbidities, history of prior procedures, preoperative pain scores, postoperative nausea, emesis, pain scores, dermatomal anesthesia, adjuvant narcotic usage, return of bowel function and length of stay (LOS).

Patients will be randomly separated into 2 groups at the time of surgery through the randomization log of the investigational drug service (IDS) pharmacy. At the request of the attending surgeon a solution will be prepared and delivered to the operating room in a blinded fashion concealed within a shielded vial.

During the abdominal component separation, dissection of the tissue planes housing the sensory fibers will be exposed to allow insertion of a large spinal needle under direct visualization on each side of the abdominal wall. Depending on the study group, the attending surgeon will inject an unknown solution (solution A or B) of either 30ml of Exparel ((bupivacaine liposome injectable suspension) 1.3% ( 13.3mg/ml)). The final test solution will be prepared in the IDS pharmacy by adding a 20 mL Exparel vial and 40cc of normal saline for a total of 60cc with a bupivacaine concentration of 0.44%. This will then be split into two 30cc solutions to be injected into each side of the transverse abdominal plane. A patient in the placebo group will be injected with 30cc of Normal Saline into the TAP region on each side of the abdomen.

All patients, independent of their study group will be provided with Patient Controlled Analgesics (PCA) using Hydromorphone or orally dosed narcotic/acetaminophen combo analgesics to ensure adequate post-operative pain control. The pain scores, dermatomal level of anesthesia, nausea, emesis, return of bowel function and length of stay will be logged into the electronic medical record. Once data collection is complete the groups will be revealed and all of the data will undergo statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects to be included are all competent patients, 18 years of age or older, who undergo abdominal component separation for a hernia.

Exclusion Criteria:

* Patients who are not having abdominal component separation or are receiving another form of regional anesthesia will be excluded.
* Patients younger than 18 years of age will be excluded.
* Amide-type local anesthetics, such as bupivacaine, are metabolized by the liver.
* Patients' with hepatic disease, because of their inability to metabolize local anesthetics normally, are at a greater risk of developing toxic plasma concentrations and will therefore be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
length of stay | participants will be followed for the duration of hospital stay, an expected average of 1 week
  determine the length of hospital stay after surgery
postoperative nausea | participants will be followed for the duration of hospital stay, an expected average of 1 week
  evaluate the presence or absence of postoperative nausea
postoperative emesis | participants will be followed for the duration of hospital stay, an expected average of 1 week
  evaluate for the presence or absence of postoperative emesis
postoperative return of bowel function | participants will be followed for the duration of hospital stay, an expected average of 1 week
  record when bowel function returns following surgery
postoperative pain score | participants will be followed for the duration of hospital stay, an expected average of 1 week
  assess pain score 0-10 a various time points following surgery

SECONDARY OUTCOMES:
adjunct narcotic pain medication use | participants will be followed for the duration of hospital stay, an expected average of 1 week
  quantify the amount of adjunct narcotic pain medication used following surgery to indirectly assess pain control obtained from the TAP block

CONTACTS AND LOCATIONS:
Overall Officials: Howard N Langstein, MD, Principal Investigator — University of Rochester Division of Plastic and Reconstructive Surgery
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Background] Girotto JA, Chiaramonte M, Menon NG, Singh N, Silverman R, Tufaro AP, Nahabedian M, Goldberg NH, Manson PN. Recalcitrant abdominal wall hernias: long-term superiority of autologous tissue repair. Plast Reconstr Surg. 2003 Jul;112(1):106-14. doi: 10.1097/01.PRS.0000066162.18720.C8. PMID 12832883
- [Background] Shestak KC, Edington HJ, Johnson RR. The separation of anatomic components technique for the reconstruction of massive midline abdominal wall defects: anatomy, surgical technique, applications, and limitations revisited. Plast Reconstr Surg. 2000 Feb;105(2):731-8; quiz 739. doi: 10.1097/00006534-200002000-00041. PMID 10697187
- [Background] Ramirez OM, Ruas E, Dellon AL. "Components separation" method for closure of abdominal-wall defects: an anatomic and clinical study. Plast Reconstr Surg. 1990 Sep;86(3):519-26. doi: 10.1097/00006534-199009000-00023. PMID 2143588
- [Background] Ewart CJ, Lankford AB, Gamboa MG. Successful closure of abdominal wall hernias using the components separation technique. Ann Plast Surg. 2003 Mar;50(3):269-73; discussion 273-4. doi: 10.1097/01.sap.0000046911.07345.0d. PMID 12800903
- [Background] Heller L, Kowalski AM, Wei C, Butler CE. Prospective, randomized, double-blind trial of local anesthetic infusion and intravenous narcotic patient-controlled anesthesia pump for pain management after free TRAM flap breast reconstruction. Plast Reconstr Surg. 2008 Oct;122(4):1010-1018. doi: 10.1097/PRS.0b013e3181858c09. PMID 18827631
- [Background] Kampe S, Warm M, Kasper SM, Diefenbach C. Concept for postoperative analgesia after pedicled TRAM flaps: continuous wound instillation with 0.2% ropivacaine via multilumen catheters. A report of two cases. Br J Plast Surg. 2003 Jul;56(5):478-83. doi: 10.1016/s0007-1226(03)00180-2. PMID 12890461
- [Background] Hivelin M, Wyniecki A, Plaud B, Marty J, Lantieri L. Ultrasound-guided bilateral transversus abdominis plane block for postoperative analgesia after breast reconstruction by DIEP flap. Plast Reconstr Surg. 2011 Jul;128(1):44-55. doi: 10.1097/PRS.0b013e3182174090. PMID 21701318
- [Background] Gorfine SR, Onel E, Patou G, Krivokapic ZV. Bupivacaine extended-release liposome injection for prolonged postsurgical analgesia in patients undergoing hemorrhoidectomy: a multicenter, randomized, double-blind, placebo-controlled trial. Dis Colon Rectum. 2011 Dec;54(12):1552-9. doi: 10.1097/DCR.0b013e318232d4c1. PMID 22067185
- [Result] Petersen PL, Mathiesen O, Torup H, Dahl JB. The transversus abdominis plane block: a valuable option for postoperative analgesia? A topical review. Acta Anaesthesiol Scand. 2010 May;54(5):529-35. doi: 10.1111/j.1399-6576.2010.02215.x. Epub 2010 Feb 17. PMID 20175754
- [Result] McDonnell JG, O'Donnell BD, Farrell T, Gough N, Tuite D, Power C, Laffey JG. Transversus abdominis plane block: a cadaveric and radiological evaluation. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):399-404. doi: 10.1016/j.rapm.2007.03.011. PMID 17961838